CLINICAL TRIAL: NCT06238193
Title: Molecular Characteristics of Early-onset Compared With Late-onset Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PRSYM202401
Record Dates: First submitted 2024-01-22; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Microsatellite Instability
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-onset colorectal cancer: Early-onset colorectal cancer
- Late-onset colorectal cancer: Late-onset colorectal cancer

SUMMARY:
The distribution rate of microsatellite instability-high (MSI-H) was significantly higher in early-onset colorectal cancer, and early-onset colorectal cancer has a specific mutational profile and relatively high programmed cell death ligand 1(PD-L1) expression, which may be used to guide personalized treatment to better control the disease.

DETAILED DESCRIPTION:
The prognosis of early-onset colorectal cancer (EOCRC) is worse than that of late-onset colorectal cancer (LOCRC), and the incidence has gradually increased in recent years, so it is necessary to study the pathogenesis and explore the target of early-onset colorectal cancer patients. In this study, investigators aimed to explore the specific molecular pathologic map of EOCRC by comparing LOCRC. This study enrolled 11,344 patients with colorectal cancer treated at the Colorectal Center of the First Affiliated Hospital of Nanjing Medical University from 2003 to 2022, of whom 578 were EOCRC and 10,766 were LOCRC. The tumor-related mutation status and tumor mutation burden (TMB) of patients were detected by next-generation sequencing technology. PD-L1 expression was detected by immunohistochemistry. The microsatellite instability was detected by polymerase chain reaction (PCR) coupled with capillary electrophoresis (2B3D NCI Panel) in all patients. Among the 11,344 patients, 180 patients with EOCRC and 90 patients with LOCRC patients underwent NGS investigation. Compared with LOCRC, EOCRC patients generally presented a later TNM stage, lower tumor differentiation, and poorer histological type. In LOCRC with MSI-H stupe, TNM stage is earlier than whom with MSI-L/MSS. In addition, the frequency of MSI-H was significantly higher in EOCRC (10.2%) than LOCRC (2.2%). The frequency of 7-mutation panel (ARID1A, FANCI, CASP8, DGFRA, DPYD, TSHR, and PRKCI) were relatively higher in LOCRC. In EOCRC group, the TNM stage of MSI-H subtype patients was earlier while harbored with worse tissue differentiation and higher proportion of mucinous adenocarcinoma. Besides, among the EOCRC patients, FBXW7, FAT1, ATM, ARID1A and KMT2B mutation frequencies were significantly increased in patients with MSI-H type. Comparing with MSI-H patients of LOCRC, the EOCRC patients with MSI-H presented a higher mutation frequencies of FGFBR2, PBRM1, RNF43, LRP1B, FBXW7, ATM and ARID1A. In addition, EOCRC patients were identified with higher tumor mutation burden, especially in the MSI-H type. PD-L1 expression calculated by tumor proportion score (TPS) was also elevated in EOCRC and correlated with MSI status.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 years old;
* Histologically proven colon or rectal adenocarcinoma.

Exclusion Criteria:

* Patients over 80 years of age;
* Recurrent colorectal cancer;
* Multiple primary tumors.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: No.
Sampling Method: Probability Sample
Enrollment: 11344 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
MSI status | Through study completion, an average of 1 year
  (I) MSI-High (MSI-H) if two or more mononucleotide markers in tumor tissue had size variations of ≥3bp compared to normal tissue; (II) MSI-Low (MSI-L) if a single mononucleotide marker in tumor tissue exhibited a size variation of ≥3bp compared to normal tissue; (III) Microsatellite Stable (MSS) if there were no size variations of ≥3bp in mononucleotide markers in tumor tissue compared to normal tissue.

SECONDARY OUTCOMES:
Copy-number variations (CNVs) | Through study completion, an average of 1 year
  Copy-number variations (CNVs) were detected using CNVkit with default parameters. Depth ratios of above 2.0(tissue) and below 0.6 were considered as CNV gain and CNV loss, respectively.

OTHER OUTCOMES:
PD-L1 level | Through study completion, an average of 1 year
  PD-L1 expression was evaluated using the Dako PD-L1 IHC 22C3 pharmDx kit (Agilent Technologies) in conjunction with the Dako Autostainer Link 48 system (Agilent Technologies). The assessment of PD-L1 expression included both the tumor proportion score (TPS) and the combined positive score (CPS).

IPD SHARING:
Plan to Share IPD: No